CLINICAL TRIAL: NCT06965517
Title: Effect of Digital Versus Static Jaw Relation Record on Crestal Bone Changes Around Implants Supporting Maxillary Single Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Lamiaa Gouda Al-Shahier B-Eid AbdelMonem Saleh, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RecID022140
Record Dates: First submitted 2025-04-15; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2023-11

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: 4 implants inserted in fully edentulous maxilla, then loading with ball abutments for maxillary overdenture
Who Masked: Outcomes Assessor
Masking Description: one of the study authors rather than the outcome assessors will take radiographic records and assess bone changes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital group (Active Comparator): implant supported maxillary overdenture constructed using electronic facebow to record maxillo-mandibular relation.
  Interventions: Procedure: Maxillary implant supported overdenture , Digital jaw relation group
- Static group (Placebo Comparator): implant supported maxillary overdenture constructed using the conventional jaw relation method
  Interventions: Procedure: Maxillary implant supported overdenture , Static jaw relation group

INTERVENTIONS:
Procedure: Maxillary implant supported overdenture , Digital jaw relation group — implant supported maxillary overdenture constructed using electronic facebow to record maxillo-mandibular relation.
  Arms: Digital group
Procedure: Maxillary implant supported overdenture , Static jaw relation group — implant supported maxillary overdenture constructed using the conventional jaw relation method.
  Arms: Static group

SUMMARY:
patients will be equally and randomly divided into 2 groups. Each group contains seven patients: Digital Group: implant supported maxillary overdenture will be constructed using electronic facebow to record maxillo-mandibular relation.

Static Group: implant supported maxillary overdenture will be constructed using the conventional jaw relation method.

Radiographic evaluation for crestal bone height around implants using direct digital periapical paralleling cone technique.

All data of radiographic evaluation were collected and tabulated then statistically analyzed using SPSS software.

DETAILED DESCRIPTION:
* Conventional single upper denture will be made for all patients.
* Occlusal adjustment of lower teeth for all patients by T-scan using the single upper conventional denture.
* The single maxillary denture will be duplicated with radiopaque markers and CBCT will be used to determine the exact positions of the implants.

Surgical procedures

1. Surgery will be done under local anesthesia.
2. Drilling will be carried out under copious sterile irrigation.
3. four implants will be inserted in canines and second premolar area in the maxilla.

After 3-4 months of implants placement, patients will be equally and randomly divided into 2 groups. Each group contains seven patients:

Digital group: For this group, implant supported maxillary overdenture will be constructed using electronic facebow to record maxillo-mandibular relation.

Static group: For this group, implant supported maxillary overdenture will be constructed using the conventional jaw relation method.

Post insertion:

* Clinical evaluation for any signs of inflammation is made.
* Further occlusal refining of lower teeth by T-scan is done with final overdenture.

Method of evaluation:

Radiographic evaluation for crestal bone height around implants using direct digital periapical paralleling cone technique.

All data of radiographic evaluation were collected and tabulated then statistically analyzed using SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Age: under 60 years.
* Completely edentulous maxillary arch.
* Opposing natural dentition in the mandibular arch.
* Residual mandibular ridge has adequate bone and covered by firm healthy mucosa.
* Class I maxillary-mandibular relationship.
* Normal salivary flow with normal viscosity.
* Systemically free patients.

Exclusion Criteria:

* Patients with poor oral hygiene.
* Patients with abnormal oral habits as (bruxism, clenching, tongue thrusting).
* Bone or mucosal diseases.
* Metabolic diseases or uncontrolled diabetes and TMJ disorders.
* Conditions that may complicate the treatment like; large tongue, gagging reflex and limited mouth opening.
* Patients who are smokers.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Marginal bone loss around implants | 18 month
  Crestal bone changes around implants supporting maxillary single overdenture opposed by natural dentition were measured using periapical radiography through long cone technique

SECONDARY OUTCOMES:
digital occlusal analysis using T-scan | 1 year
  Immediately after implant overdenture insertion, occlusal force magnitude, time and equilibrium were measured by the T-scan digital system by instructing the patient to bite on a sensor attached to a laptop on which the biting force was displayed as a count of disocclusion time and occlusion time, dictating the degree of any occlusal interference. The system also shows the degree of centralization of biting force between the right and left sides of the arch.

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa GA Saleh, BSc, MSc, Principal Investigator — Faculty of Dentistry, Ain Shams University
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
a data availability statement will be provided in the article going to be published indicating that data will be available upon reasonable request from the principle investigator
Supporting Information: Study Protocol, SAP
Time Frame: the data will become available along with publishing the article